CLINICAL TRIAL: NCT04655248
Title: ACURATE neo2™ Post Market Clinical Follow up Study
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2410
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Calcification; Aortic Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Aortic Diseases | interventions — Transcatheter Aortic Valve Replacement; Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation/Replacement — The device is placed in patients heart at the level of aortic valve through a transfemoral access from femoral groin as indicated in device IFU

SUMMARY:
The ACURATE Neo2 PMCF is aimed at collecting clinical and device performance outcomes data with the ACURATE neo2™ Transfemoral Aortic Valve System as used in routine clinical practice for the treatment of severe calcific aortic stenosis.

DETAILED DESCRIPTION:
ACURATE neo2 PMCF is a prospective, open-label, single-arm, multicenter, observational post-market surveillance study. All subjects deemed treatable with the ACURATE neo2 valve will be approached to participate in the study.

A subject who provides an Informed Consent Form (ICF) approved by the Independent Ethics Committee (IEC) and signed by the subject or the subject's legally authorized representative is considered enrolled once an attempt is made to insert the commercially available ACURATE neo2 Transfemoral Delivery System. Approximately 200 subjects will be enrolled.

Follow-up will occur at pre-discharge, 30 days, 1 year, and then annually from 2 through 5 years post index procedure per standard of care. Visits are in-person through 1 year and in-person (preferred) or via telephone interview in years 2 through 5. All subjects will undergo 4D computed tomography (CT) imaging at 30 days and 1 year.

ACURATE neo2 PMCF Study Design Overview Abbreviations: CT=computed tomography; ICF=Informed Consent Form

ELIGIBILITY:
Inclusion Criteria:

There are no specific inclusion criteria set for this post-market surveillance study. A subject must sign an IEC-approved ICF and the ACURATE neo2 Transfemoral Aortic Valve System should be used according to the commercial IFU.

Exclusion Criteria:

EC1. Subject has a previous bioprosthesis in the aortic position.

EC2. Subject has eGFR <30 mL/min (chronic kidney disease stage IV or stage V).

EC3. Subject has atrial fibrillation that cannot be rate controlled to ventricular response rate < 60 bpm.

EC4. Subject is expected to undergo chronic anticoagulation therapy after the TAVI procedure

Note : Subjects treated with short-term anticoagulation post-procedure can be included; in these subjects the 30-day imaging will be performed 30 days after discontinuation of anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic heart disease due to severe native calcific aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: | 30 days
  All-cause mortality after the index implant procedure
Primary Imaging Endpoint: | 30 days
  Hypoattenuated leaflet thickening (HALT) as measured by 4D CT

SECONDARY OUTCOMES:
Safety endpoints adjudicated by an independent Clinical Events Committee | all 5 years
  All-cause mortality (cardiovascular and non-cardiovascular) Stroke (disabling and non-disabling) Bleeding (life-threatening [or disabling] and major) Vascular complications (major) Hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV)
Additional Safety Endpoints | all 5 years
  * Myocardial infarction (periprocedural [≤72 hours post index procedure] and spontaneous [>72 hours post index procedure])
  * Acute kidney injury (≤7 days post index procedure) based on the AKIN System Stage 3 (including renal replacement therapy) and Stage 2
  * Repeat procedure for valve-related dysfunction (surgical or interventional therapy)
  * New permanent pacemaker implantation resulting from new or worsened conduction disturbances
  * New onset of atrial fibrillation or atrial flutter
  * Coronary obstruction (≤3 days post index procedure)
  * Ventricular septal perforation (≤3 days post index procedure)
  * Annular rupture (≤3 days post index procedure)
  * Cardiac tamponade (≤3 days post index procedure)
  * Valve migration
  * Valve embolization
  * Ectopic valve deployment
  * Transcatheter aortic valve (TAV)-in-TAV deployment
  * Prosthetic aortic valve thrombosis
  * Prosthetic aortic valve endocarditis
Prosthetic Aortic Valve Performance as measured by transthoracic echocardiography (TTE) | Discharge, 30 days, annually from year 1 to 5
  Effective orifice area (EOA), Mean and Peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation/paravalvular leak (PVL).
  Center-reported TTE measures will also be collected annually at 2 through 5 years per local standard of care for TAVI.
EuroQoL Quality of Life questionnaire (EQ-5D-5L) | Baseline, 30-day, 1-year
  Health status as evaluated by the EQ-5D-5L Quality Of Life questionnaire
New York Heart Association (NYHA) functional classification | Baseline, Discharge, 30 days, annually from year 1 to 5
  Classification of heart failure symptoms as evaluated by NYHA classification
Assessments using 4D CT-scan | 30 days 1 year
  * Assessment of leaflet mobility
  * Assessment of hypoattenuated leaflet thickening (HALT)
  * Assessment of leaflet thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Won-Keun Kim, MD, Principal Investigator — Kerckhoff Klinik
Locations (19):
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Germany (4):
  - Kerckhoff-Klinik GmbH Herz und Thorax Zentrum Abteilung Kardiologie/Kardiochirurgie, Bad Nauheim
  - HDZ Bad Oeynhausen, Bad Oeynhausen
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinik Regensburg, Regensburg
- Italy (3):
  - A.O.U Policlinico "G.Rodolico - San Marco", Catania, CA
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliera Pisana, Pisa
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht, Utrecht
- Spain (2):
  - Hospital Clinico de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario Valladolid, Valladolid
- Sweden (2):
  - Lund University, Cardiology department, Lund
  - Karolinska Universitetssjukhuset, Stockholm
- Universitätsspital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy. (http://www.bostonscientific.com/en-US/data-sharing-requests.html)

REFERENCES:
- [Derived] Kim WK, Mollmann H, Montorfano M, Ellert-Gregersen J, Rudolph TK, Van Mieghem NM, Hilker M, Amat-Santos I, Terkelsen CJ, Petronio AS, Stella P, Gotberg M, Ruck A, Kasel AM, Trillo R, Appleby C, Barbanti M, Blanke P, Asch FM, Modolo R, Allocco DJ, Tamburino C. Outcomes and performance of the ACURATE neo2 transcatheter heart valve in clinical practice: one-yearresults of the ACURATE neo2 PMCF Study. EuroIntervention. 2024 Jan 1;20(1):85-94. doi: 10.4244/EIJ-D-23-00823. PMID 37982152